CLINICAL TRIAL: NCT03318419
Title: Efficacy and Safety of Cladribine in Combination With G-CSF, Low-dose Cytarabine and Pegaspargase in Patients With Refractory/Relapsed Acute Lymphoblastic Leukemia: a Phase 2 Clinical Trial
Brief Title: Cladribine in Combination With GAP in Patients With Refractory/Relapsed Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, dr. luyue, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALL-2017
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cladribine; Granulocyte Colony-Stimulating Factor; Cytarabine; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cladribine group (Experimental): Cladribine in combination of GAP (G-CSF priming, low dose cytarabine, and Pegaspargase) will be administrated in this arm
  Interventions: Drug: Cladribine; Drug: G-CSF; Drug: Cytarabine; Drug: Pegaspargase

INTERVENTIONS:
Drug: Cladribine — 5mg/㎡ d1-5
  Other Names: cladribine injection
Drug: G-CSF — 300ug d0-14
  Other Names: granulocyte
Drug: Cytarabine — 10mg/㎡ q12h SC d1-14
  Other Names: Ara-C
Drug: Pegaspargase — 2500U/m2 im d1
  Other Names: Pegaspargase injection

SUMMARY:
The vast majority of patients with ALL will die of the disease, and no standard chemotherapy regimen were defined for patients with relapsed/refractory ALL.Our previous experience has shown that Cladribine in combination of GAP (G-CSF priming, low dose cytarabine, and Pegaspargase) are effective with tolerable toxicity profiling.Thus, this phase 2 clincial trial is going to evaluate the efficacy and safety of cladribine in combination with G-CSF, low-dose cytarabine and Pegaspargase (C-GAP) in patients with refractory/relapsed acute Lymphoblastic Leukemia

DETAILED DESCRIPTION:
ALL is common in the elderly patients, who can not tolerate the intensified treatments. The vast majority of patients with ALL will die of the disease, and no standard chemotherapy regimen were defined for patients with relapsed/refractory ALL. Our previous experience has shown that Cladribine in combination of GAP(G-CSF priming, low dose cytarabine, and Pegaspargase) are effective with tolerable toxicity profiling.Thus, this phase 2 clincial trial is going to evaluate the efficacy and safety of cladribine in combination with G-CSF, low-dose cytarabine and aclarubicin (C-CAG) in patients with refractory/relapsed acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* Clinical diagnosis of Relapsed/Refractory ALL;
* ECOG performance status (PS) score 0-3;
* AST and ALT <=2.5 times the institutional ULN;
* Total bilirubin <=2.0 times the institutional ULN
* Serum creatinine<2.0 times the institutional ULN;
* Subjects should take effective contraceptive measures，and serum or urine pregnancy tests must be negative during the screening and study periods in women subjects;
* Patients should understand the disease and voluntarily receive the study regimen and follow-up.

Exclusion Criteria:

* Concurrent diagnosis of tumors other than ALL, with exclusion of superficial bladder cancer, basal cell and squamous cell carcinoma, cervical intraepithelial neoplasms (CIN), prostatic intraepithelial neoplasms(PIN);
* Active viral or bacterial infection that would impair the ability of the subject to receive protocol therapy;
* Concurrent autoimmune hemolytic anemia or immune thrombocytopenia;
* Subjects suffered from AIDS，active hepatitis B or C virus infection;
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent;
* Be allergic to any component of C-GAP regimen;
* Subjects ever exposed to cladribine or CAG-based regimen.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
CR rate | Bone marrow aspiration will be done within 2 weeks after blood cell count recovery (about 4 weeks after initiation of C-GAP treatment
  Complete Remission: less than 5% blasts in bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: yue lv, MD., Principal Investigator — sun-yat sun university cancer center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No